CLINICAL TRIAL: NCT06954298
Title: Metabolic Dysregulation as the Underlying Principle of Integrated Pathophysiology of Obesity-associated Chronic Diseases: Molecular Landscape of Complex Lifestyle Modification
Brief Title: Molecular Landscape of Complex Lifestyle Modification
Acronym: COPMose
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: Medical University Vienna (Unknown)
Responsible Party: Principal Investigator, Jozef Ukropec, PhD, DSc, Slovak Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 09I03-03-V04-00555
Record Dates: First submitted 2025-03-30; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obesity Prevention; Obesity; Metabolic Disease
Keywords: lifestyle intervention; exerkines; metabolic flexibility
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lifestyle intervention (Experimental)
  Interventions: Behavioral: supervised lifestyle modification
- Control (No Intervention)

INTERVENTIONS:
Behavioral: supervised lifestyle modification — Supervised lifestyle intervention will consist of regular exercise (3x a week), nutritional counselling (weekly), cognitive bahavioural therapy (monthly).
  Arms: lifestyle intervention

SUMMARY:
The goal of this clinical trial is to detect the impact of the 3-month complex lifestyle intervention, consisting of dietary counselling, supervised exercise training and cognitive-behavioural intervention in middle-aged sedentary individuals with obesity, specific questions are:

* What is the adaptive response to exercise training on the whole-body and skeletal muscle energy metabolism, insulin sensitivity, metabolic flexibility, muscle functional parameters and cardiopulmonary fitness?
* Would the intensity-related changes of the exercise-induced substrate preference (lipids vs carbohydrates) be a good predictive marker of metabolic flexibility i.e. the capacity to reduce the whole-body metabolic burden in patients with obesity?
* Is the signal driving the adaptive response to regular exercise contained in serum derived Extracellular vesicles?

Researchers will examine effects of exercise training intervention on whole body energy metabolism, by integrating clinical, biochemical and molecular data.

Participants will:

* Undergo 3 months exercise - intervention program.
* Be submitted to examination of their obesity, energy metabolism and cardiopulmonary fitness related phenotypes using bioelectric impedance, indirect calorimetry, cycle spiroergometry.
* Blood samples will be taken both, at the baseline PRE- and POST- intervention.

ELIGIBILITY:
Inclusion Criteria: BMI 30-45 kg.m-2 -

Exclusion Criteria: smoking, cancer,

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic flexibility in response to submaximal exercise and nutritional challenge | 24 months
  Metabolic flexibility (metabolic substrate switching) will be measured using indirect calorimetry during submaximal exercise test (on stationary bike) and in response to nutritional challenge (fasting / glucose uptake during oGTT)

SECONDARY OUTCOMES:
cardiopulmonary fitness (VO2max) | 24 months
  Cardiopulmonary fitness will be measured by bicycle spiro-ergometry
Index of insulin resistance (oGTT) | 24 months
  Index of insulin resistance will be calculated from the results of the frequently sampled oral glucose tolerance test oGTT.
abdominal adiposity and abdominal adipose tissue distribution (subcutaneous / visceral) | 24 months
  abdominal adiposity will be assessed by quadrupedal biopimpedance, and adipose tissue distribution by magnetic resonance imagining

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ukropcová, Prof. MD PhD, Study Chair — Biomedical Research Center Slovak Acad Sci; Jozef Ukropec, PhD, DSc, Principal Investigator — Biomedical Research Center Slovak Acad Sci
Locations (1):
- Center for Obesity Management EASO, Biomedical Research Center SAS, Bratislava, Bratislava Region, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and SAP will be available upon study completion, and primary and secondary outcomes (clinical study report) will be shared after publishing the results in a scientific journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 06/2026 (start date) indefinitely (end date)
Access Criteria: researchers with legitimate interest